CLINICAL TRIAL: NCT05490082
Title: Mirabegron, Propevirine, Solifenacin for Treatment of Lower Urinary Tract Symptoms During Intravesical BCG Instillation: Prospective Randomized Controlled Trial
Brief Title: Mirabegron, Propevirine, Solifenacin for Treatment of Lower Urinary Tract Symptoms During Intravesical BCG Instillation
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ali Elmenair, principle investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MD.21.12.576
Record Dates: First submitted 2022-06-30; First posted 2022-08-05 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Voiding Disorders
MeSH Terms: interventions — mirabegron; Solifenacin Succinate

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mirabegron arm (Active Comparator): 50 mg PO once daily
  Interventions: Drug: Mirabegron, Propevirine, Solifenacin
- Propevirine arm (Active Comparator): 15 mg PO twice daily
  Interventions: Drug: Mirabegron, Propevirine, Solifenacin
- Solifenacin arm (Active Comparator): 10 mg PO once daily
  Interventions: Drug: Mirabegron, Propevirine, Solifenacin
- Placebo arm (Placebo Comparator): starch tablet once daily
  Interventions: Drug: Mirabegron, Propevirine, Solifenacin

INTERVENTIONS:
Drug: Mirabegron, Propevirine, Solifenacin — Efficacy comparison

SUMMARY:
A randomized controlled study to compare the efficacy of mirabegron, solifenacin and propevirine for treatment of Lower urinary tract symptoms during intravesical BCG installation

ELIGIBILITY:
Inclusion Criteria:

* Patients older than age 18 years.
* Able to provide an informed consent.
* Denovo or recurrent cases with intermediate and high risk NMIBC eligible for intravesical BCG immunotherapy.
* Persistent LUTS after intravesical BCG induction.

Exclusion Criteria:

* International Prostate symptom score (IPSS) greater than 20.
* Post-void residual (PVR) volume greater than 50 ml.
* Use of medications for overactive bladder.
* Pelvic surgery within the previous 6 months.
* Hypersensitivity for BCG or any of the above mentioned drugs.
* Tumor recurrence during follow up period.
* Other medical conditions that would be adversely affected by anticholinergics such as history of urinary retention due to BPH(Benign prostatic hyperplasia), constipation and history of narrow angle glaucoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Dysuria | 3 months
  Compare the percentage of reduction of dysuria as measured by Pain Visual Analouge Score at 3 month follow up after using propiverine, mirabegron and solifenacin versus placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Elhefnawy, MD, Study Director — Urology and Nephrology Center Mansoura University
Locations (1):
- Urology and Nephrology Center, Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No